CLINICAL TRIAL: NCT00918970
Title: Interest of Real Time Measurement of Autonomous Nervous System for the Detection of Brain Death: the MEANS Study
Brief Title: Interest of Real Time Measurement of Autonomous Nervous System for the Detection of Brain Death
Acronym: MEANS
Status: Terminated | Type: Observational
Why Stopped: Angioscanners in excess of the SNA group because of use of thiopental
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: David CHARIER, CHU de SAINT-ETIENNE
Other Study IDs: 0708045; CNIL 908.476
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Cerebral Hematoma, Traumatic; Intracerebral Hemorrhage, Traumatic; Traumatic Brain Hemorrhage; Traumatic Brain Injury
Keywords: autonomous nervous system; brain death; organs transplantation
MeSH Terms: conditions — Cerebral Hemorrhage, Traumatic; Brain Hemorrhage, Traumatic; Brain Injuries, Traumatic; Brain Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SNA group: This group will have a real-time analysis of autonomic nervous system activity during its intensive care hospitalisation
- Clinical group: This group will have a conventional clinical analysis during its intensive care hospitalisation

SUMMARY:
Context: A major lack of organ donors is a serious public health problem. It determines a prolonged delay before a transplant can be performed and thus a significant number of deaths of patients waiting for transplantation. The aim of this project is to reduce the delay of the diagnosis of brain death, and also to improve its diagnosis in the Intensive Care Unit.

The diagnosis of brain death is strictly defined by the law and relies either on two consecutive flat electroencephalograms recorded at an interval of four hours, or on the lack of cerebral circulation during a brain angiography performed after suspecting brain death on the clinical exam. However, in usual practice, it is difficult to have all the needed clinical arguments, and their interpretation can be difficult in the pathological context. This may participate in the delay and the lack of patients potentially donors.

Pre-study: In a pilot study, fifty subjects with severe cerebral lesions, had a continuous ECG recording. The investigators could find that a decrease in autonomic nervous system activity, as measured through the ECG, was correlated to the transition to brain death assessed by cerebral angiography. The loss of cardiac variability was always observed between two cerebral angiographies, one before and the second after brain death. This study allowed the investigators to calculate the threshold values of sympathetic and parasympathetic activities to confirm brain death.

DETAILED DESCRIPTION:
Aim: The aim of this second study is to validate prospectively the interest of the analysis in real-time of autonomic nervous system activity to detect brain death.

Benefits expected: Increase the number of organ donors and the number of organs removal available for transplantation.

ELIGIBILITY:
Inclusion Criteria:

* severe cerebral lesions
* admitted in intensive care units

Exclusion Criteria:

* neoplastic pathology
* prior myocardiac infarction
* hearth failure
* atrial fibrillation
* insulin-treated diabetes mellitus
* cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with severe cerebral lesions admitted in intensive care units
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
the delay between the falling down of autonomic nervous system activity and the confirmation of the brain death using cerebral angiography | At confirmation of the brain death

SECONDARY OUTCOMES:
the number of patients and the number of organs removed | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: David CHARIER, MD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - CHU de Dijon, Dijon
  - CH Roanne, Roanne
  - CHU de Saint-Etienne, Saint-Etienne